CLINICAL TRIAL: NCT02327260
Title: Increasing Adherence to Treatment Recommendations Following a Cardiac Event
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Kymberley Bennett, Associate Professor, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-521
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Videotape Recording; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Video + MI for CR (Experimental): This group receives the educational video and an MI session for CR participation.
  Interventions: Behavioral: Video + Motivational interview for CR participation
- MI for medication adherence (Experimental): This group receives an MI session for taking prescribed cardioprotective medications.
  Interventions: Behavioral: Motivational interview for medication adherence
- Control group (standard care) (No Intervention): The control group receives standard care while hospitalized.

INTERVENTIONS:
Behavioral: Video + Motivational interview for CR participation — Patients will be shown a 9 minute video that highlights actual CR patients discussing barriers they overcame to participate in CR, and introductions to the CR staff. The brief, phone-based motivational interview will focus on increasing motivation to participate in CR.
  Arms: Video + MI for CR
Behavioral: Motivational interview for medication adherence — The brief, phone-based motivational interview will focus on increasing motivation to adhere to prescribed cardioprotective medications.
  Arms: MI for medication adherence

SUMMARY:
This project will pilot test an intervention to increase participation rates in cardiac rehabilitation and medication adherence among patients following a cardiovascular event. The intervention will use an educational video shown during referral to cardiac rehabilitation (before hospital discharge), along with a brief, telephone-delivered counseling session to increase motivation to participate in cardiac rehabilitation and take all cardiac medications as prescribed (following hospital discharge). One hundred twenty patients who have experienced a cardiovascular event, and who are eligible for cardiac rehabilitation, will be recruited to participate in the study. Three groups of participants (40 each) will be formed: a control group that receives standard care, a first experimental group that sees the educational video and receives motivational counseling to attend cardiac rehabilitation, and a second experimental group that receives motivational counseling to adhere to their medications as prescribed. It is expected that the experimental group participants will differ from the control group participants in rates of participation in cardiac rehabilitation (experimental group #1) and medication adherence (experimental group #2). If successful, this intervention could be used in hospital settings to increase patients' adherence behaviors.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of a pilot intervention to increase adherence behaviors among patients eligible for cardiac rehabilitation (CR). The intervention will include two components. The first component is an educational video shown pre-discharge, at the time referral to CR is made. The video, based on social-cognitive principles, will educate patients about what they can expect during CR using actual CR patients. The second component of the intervention will be a brief, telephone-delivered counseling session to increase motivation to adhere to prescribed CR participation or cardiac medications. The counseling session will use well-established motivational interviewing techniques. Three groups will be formed, with 40 participants each: a control group that receives standard care, experimental group #1 that receives the educational video plus a counseling session that focuses on participating in CR, and experimental group #2 that receives a counseling session that focuses on taking cardiac medications as prescribed.

Given that this is a pilot study and the sample size is relatively small, statistically significant differences are not expected. However, the following hypotheses will be explored:

* Experimental group #1 will differ from the control group in rates of participation in CR.
* Experimental group #2 will differ from the control group and experimental group #1 in adherence to prescribed medications.

Participants will be recruited from patients at Truman Medical Center (TMC) who are eligible for CR. Information is received daily about new patients at TMC who are eligible for CR and who need to be referred. Investigators will provide research team members information about eligible patients who can be approached about study participation. A member of the research team will visit patients in their TMC hospital rooms pre-discharge and ask if they are interested in learning about the study. If they indicate an interest in learning more, a brief summary of the study will be provided (e.g., "The investigators are interested in learning about how health care providers can best talk to patients about treatment recommendations."). Then, the team member will administer a brief cognitive assessment to determine whether the patient is able to complete the study to determine if inclusion criteria are met. If they decline participation, or if they do not correctly answer the first two screening questions, patients will be asked to answer five brief demographic questions and thanked for their time. These five demographic questions will be asked so that investigators may compare the final sample to patients who declined participation to explore for differences that could limit generalizability of findings.

If a patient correctly answers the two screening questions, and continues to be interested in learning more about the study, the research team member will provide the patient with a consent form and TMC's PHI authorization form. Upon completion of the consent form, patients also will be asked to review the pharmacy release form and complete and sign it if they consent to sharing their prescription refill data with investigators. Afterward, the Time 1 (baseline) questionnaire will be administered via interview by the research team member. The interview will take approximately 15 minutes to complete. Upon completion, the research team member will provide the participant with an appointment reminder card and a $10 cash voucher than can be used at the TMC Cash Office. At that time, the team member will schedule the next two interviews to be completed by telephone (i.e., Times 2 and 3).

Upon completion of the Time 1 questionnaire, the team member will complete a form with the participant's basic information and provide it to the CR nurse. In turn, the CR nurse will assign the participant to one of the three study groups. Before recruitment begins, a statistician will create a random number table with group assignments stratified by race and heart failure diagnosis. The random number table will be used to create sealed envelopes with randomization information for each study participant. The envelopes will be sequentially numbered and provided to the CR nurse before recruitment. Upon receiving a form from a team member, she will open the next sealed envelope to reveal into which group the participant is assigned. She will note the envelope number and group assignment on the form. Then, the form will be provided to the research team for secure storage.

Participants will be randomly assigned to one of three groups:

A control group that receives standard care. Standard care includes a visit by the CR nurse pre-discharge to refer the patient to CR. This referral session includes a discussion of heart health, CR benefits and outcomes, and literature about prescribed medications. If possible, the CR orientation appointment is scheduled with patients. If it is not possible to schedule the orientation session at the referral, CR staff members call the patient a few days after discharge to schedule an appointment. Reminder calls are made by CR staff members a few days before scheduled appointments. The pharmacist also visits all patients after the CR referral is made to review prescribed medications. Follow-up phone calls are made 2-3 days after discharge by the pharmacy team to answer any medication questions and trouble-shoot any problems.

Experimental group #1: This group will receive standard care (detailed above), and it will be shown the educational video on an iPad by the CR nurse during referral. The educational video will be based on social-cognitive principles, with the goal of educating prospective CR patients about what happens during CR. The video will be approximately nine minutes long, and will feature testimonials by real CR patients. In addition, this group will be called by a trained counselor approximately one week after discharge. During this call, the counselor will conduct a brief counseling session, using motivational interviewing (MI) techniques, that focuses on increasing motivation to participate in CR. During this session, the counselor will help the participant identify barriers and benefits to participating in CR, thereby increasing internal motivation to participate. The counseling session will take approximately 10 minutes.

Experimental group #2: This group will receive standard care (detailed above), plus a counseling session that focuses on medical adherence. Specifically, the counselor will conduct a session on improving internal motivation to adhere to the cardiac medications prescribed by the pharmacist. The session will take approximately 10 minutes.

As stated above, the CR nurse will note the participant's randomization on the information sheet, and this information will be shared with the other research team members after the participant is discharged from the hospital. This information will be shared with team members prior to the Time 2 phone call (because group membership needs to be determined before the call is made to plan for which, if any, counseling session will be completed).

All participants will take part in the Time 1 interview (see above), as well as telephone interviews at Time 2 (approximately one week post-discharge; immediately prior to the counseling session provided to the experimental groups) and Time 3 (approximately five weeks post-discharge). The Time 2 interview will take approximately 20 minutes and the Time 3 interview will take approximately 30 minutes.

Therefore, the control group will take part in a 15-minute Time 1 in-person interview, a 20-minute Time 2 telephone interview, and a 30-minute Time 3 telephone interview. Experimental group #1 will take part in a 15-minute Time 1 in-person interview, a 20-minute Time 2 telephone interview, a 10 minute counseling session immediately following the Time 2 interview, and a 30-minute Time 3 telephone interview. Experimental group #3 will take part in a 15-minute Time 1 in-person interview, a 20-minute Time 2 telephone interview, a 10-minute counseling session immediately following the Time 2 interview, and a 30-minute Time 3 telephone interview.

The Time 1 (baseline) interview measures the following constructs/contains the following scales:

* Demographic questions
* Confidence and motivation to change behaviors
* Knowledge about cardiac rehabilitation
* Patient Health Questionnaire (PHQ-9)
* Perceived Stress Scale (PSS)
* Subjective health status (adapted from BRFSS)
* Cardiac self-blame

The Time 2 (1-week post-discharge) interview measures the following constructs/contains the following scales:

* Confidence and motivation to change behaviors
* Medication Adherence Self-Efficacy
* Treatment Self-Regulation Questionnaire
* Knowledge about cardiac rehabilitation
* Knowledge about cardioprotective medications
* Patient Health Questionnaire (PHQ-9)
* Perceived Stress Scale (PSS)
* Subjective health status (adapted from BRFSS)
* Medical Care Questionnaire
* Medication Adherence
* Feedback about educational video (not for control/experimental group #2)

The Time 3 (5-weeks post-discharge) interview measures the following constructs/contains the following scales:

* Confidence and motivation to change behaviors
* Medication Adherence Self-Efficacy
* Treatment Self-Regulation Questionnaire
* Knowledge about cardiac rehabilitation
* Knowledge about cardioprotective medications
* Patient Health Questionnaire (PHQ-9)
* Perceived Stress Scale (PSS)
* Subjective health status (adapted from BRFSS)
* Medical Care Questionnaire
* Medication Adherence
* Ratings of the counseling session (not for control group)

ELIGIBILITY:
Inclusion Criteria:

1. Referral to CR according to the AACVPR/ACCF/AHA guidelines
2. English speaking
3. At least 18 years of age
4. Lack of physical or cognitive impairments that would limit patients' abilities to complete study materials or participate in CR.

Exclusion Criteria:

1. Physical impairment such as debilitating stroke or another medical condition that would limit their ability to complete the study materials or participate in CR
2. Patients transferred to an outside facility for revascularization procedures
3. Previous participation in this research protocol (i.e. patients can only participate one time)
4. Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Truman Medical Center, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited for the study between March 2015 and May 2016. Patients were approached for study inclusion during hospitalization following a cardiac procedure.
Groups:
- MI for Medication Adherence: This group receives an MI session for taking prescribed cardioprotective medications,
  Motivational interview for medication adherence: The brief, phone-based motivational interview will focus on increasing motivation to adhere to prescribed cardioprotective medications.
- Control Group (Standard Care): This is the standard of care group. It received typical care by hospital staff following a cardiac procedure.
Period: Overall Study
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Started | 20 | 24 | 17
Completed | 14 | 20 | 15
Not Completed | 6 | 4 | 2
Not completed — Lost to Follow-up | 2 | 3 | 2
Not completed — invalid phone number | 1 | 1 | 0
Not completed — non-adherence to protocol | 2 | 0 | 0
Not completed — cognitive concerns | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group (Standard Care): This group received standard care following a cardiac procedure.
- Total: Total of all reporting groups
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care) | Total
Number analyzed (Participants) | 14 | 20 | 15 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.50 (8.71) | 57.50 (7.96) | 55.93 (7.06) | 56.45 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 4 | 17
  Male | 9 | 12 | 11 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 3 | 16
  White | 8 | 11 | 12 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 20 | 15 | 49

OUTCOME MEASURES:

1. Primary Outcome: Participation in CR
Description: Whether participants attend an orientation session at TMC's CR program
Time Frame: Within 2 months of study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 14 | 20 | 15
Participants | 7 | 11 | 6

2. Primary Outcome: Adherence (Ratio): P2Y12 Platelet Inhibitor
Description: A continuous single-interval medication availability ratio was calculated by dividing the number of days supplied by a pharmacy fill by the number of days before the next pharmacy fill for the same medication. A higher ratio was indicative of greater adherence.
Time Frame: Collected at 5 weeks post-discharge
Population: Some pharmacies did not respond to us after repeated requests for participants' data; therefore, data are missing.
Measure: Mean (Standard Deviation); unit: adherence ratio
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 12 | 15 | 9
adherence ratio | .47 (.44) | .72 (.44) | .46 (.46)

3. Primary Outcome: Adherence (Ratio): Beta-Blocker
Description: as for outcome 2
Time Frame: Collected at 5 weeks post-discharge
Population: We are missing data because some pharmacies did not respond to our requests.
Measure: Mean (Standard Deviation); unit: adherence ratio
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 12 | 15 | 9
adherence ratio | .20 (.36) | .39 (.49) | .40 (.48)

4. Primary Outcome: Adherence (Ratio): Statin
Description: as for outcome 2
Time Frame: Collected at 5 weeks post-discharge
Population: We are missing data because some pharmacies did not respond to our requests.
Measure: Mean (Standard Deviation); unit: adherence ratio
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 12 | 15 | 9
adherence ratio | .22 (.44) | .37 (.48) | .46 (.45)

5. Primary Outcome: Adherence (Ratio): Angiotensin System Blocker
Description: as for outcome 2
Time Frame: Collected at 5 weeks post-discharge
Population: We are missing some data because pharmacies did not respond to our requests.
Measure: Mean (Standard Deviation); unit: adherence ratio
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 12 | 15 | 9
adherence ratio | .26 (.43) | .44 (.53) | .91 (.13)

6. Primary Outcome: Number of Participants With Self-reported Medication Adherence: P2Y12 Platelet Inhibitor
Description: Participants were asked how many times they filled P2Y12 Platelet Inhibitors since their discharge from TMC. Participants were coded as "adherent" if they reported an increased number of medication fills at 5 weeks compared to 1 week post-discharge. Participants with evidence of obtaining a medication fill greater than 30 days were also classified as "adherent." Participants who did not indicate an increase in number of fills or provide evidence of extended coverage from initial fill were determined to be "non-adherent." Dichotomized adherence categorization was utilized in data analyses: 1 = adherent; 0 = non-adherent. Data presented are % adherent.
Time Frame: Interview data at 5 weeks post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 14 | 20 | 15
Participants | 9 | 5 | 7

7. Primary Outcome: Number of Participants With Self-reported Medication Adherence: Beta-Blocker
Description: Participants were asked how many times they filled Beta-Blockers since their discharge from TMC. Participants were coded as "adherent" if they reported an increased number of medication fills at 5 weeks compared to 1 week post-discharge. Participants with evidence of obtaining a medication fill greater than 30 days were also classified as "adherent." Participants who did not indicate an increase in number of fills or provide evidence of extended coverage from initial fill were determined to be "non-adherent." Dichotomized adherence categorization was utilized in data analyses: 1 = adherent; 0 = non-adherent. Data presented are % adherent.
Time Frame: Interview data at 5 weeks post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 14 | 20 | 15
Participants | 10 | 8 | 8

8. Primary Outcome: Number of Participants With Self-reported Medication Adherence: Statin
Description: Participants were asked how many times they filled Statins since their discharge from TMC. Participants were coded as "adherent" if they reported an increased number of medication fills at 5 weeks compared to 1 week post-discharge. Participants with evidence of obtaining a medication fill greater than 30 days were also classified as "adherent." Participants who did not indicate an increase in number of fills or provide evidence of extended coverage from initial fill were determined to be "non-adherent." Dichotomized adherence categorization was utilized in data analyses: 1 = adherent; 0 = non-adherent. Data presented are % adherent.
Time Frame: Interview data at 5 weeks post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 14 | 20 | 15
Participants | 10 | 9 | 12

9. Primary Outcome: Number of Participants With Self-reported Medication Adherence: Angiotensin System Blocker
Description: Participants were asked how many times they filled Angiotensin System Blockers since their discharge from TMC. Participants were coded as "adherent" if they reported an increased number of medication fills at 5 weeks compared to 1 week post-discharge. Participants with evidence of obtaining a medication fill greater than 30 days were also classified as "adherent." Participants who did not indicate an increase in number of fills or provide evidence of extended coverage from initial fill were determined to be "non-adherent." Dichotomized adherence categorization was utilized in data analyses: 1 = adherent; 0 = non-adherent. Data presented are % adherent.
Time Frame: Interview data at 5 weeks post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
Number analyzed (Participants) | 14 | 20 | 15
Participants | 11 | 11 | 7

ADVERSE EVENTS:
Description: Adverse events were not assessed because none was anticipated given the focus of the study.
Arm/Group | Video + MI for CR | MI for Medication Adherence | Control Group (Standard Care)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes